CLINICAL TRIAL: NCT03377387
Title: Phase Ib/II Study of Capecitabine 7/7 Schedule With Neratinib in Patients With Metastatic HER2-Positive Breast Cancer
Brief Title: Capecitabine 7/7 Schedule With Neratinib in Patients With Metastatic HER2-Positive Breast Cancer
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Puma Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-585
Record Dates: First submitted 2017-12-14; First posted 2017-12-19 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer
Keywords: Capecitabine; Neratinib; HER2-Positive; 17-585
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine; neratinib

STUDY DESIGN:
Intervention Model Description: This is a phase Ib/II study of capecitabine 7/7 with neratinib in patients with HER2-positive metastatic breast cancer.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- capecitabine 7/7 with neratinib (Experimental): In the phase I portion of the study, a 3+3 design will be used. Once the MTD is reached, the phase II portion will enroll up to 24 patients. Capecitabine will be taken orally in AM and PM (at the assigned dose per cohort) 7 days on and 7 days off. Neratinib is given as 240 mg daily continuously without stopping. A cycle is 28 days. Patients will be seen on Day 1 of each cycle (+/- 3 days).
  The MD has been determined as 240mg of neratinib and 1000mg BID of capecitabine.
  Interventions: Drug: Capecitabine; Drug: Neratinib; Behavioral: EORTC QLQ - BR23, EQ-5D-5L, EORTC QLQ-C30

INTERVENTIONS:
Drug: Capecitabine — Capecitabine will be taken orally in AM and PM (at the assigned dose per cohort) 7 days on and 7 days off. Phase II MD 1000mg BID of capecitabine.
Drug: Neratinib — Neratinib is given as 240 mg daily continuously without stopping. A cycle is 28 days. Phase II The MD has been determined as 240mg of neratinib
Behavioral: EORTC QLQ - BR23, EQ-5D-5L, EORTC QLQ-C30 — Questionnaires Every Cycle (+/- 3 days) (For phase II)

SUMMARY:
This is a phase l/II study. The purpose of this study is to test the safety of the study drug neratinib in combination with a standard chemotherapy drug called capecitabine at different doses to find out what effects, if any, it has on people. Capecitabine (Xeloda®) is approved by the Food and Drug Administration (FDA) for advanced breast cancer treatment. Neratinib is an investigational drug, meaning the FDA has not approved the use of this drug for advanced breast cancer. The combination of capecitabine and neratinib has been studied before in another study where capecitabine was administered using the standard dosing schedule. In this study, the investigators want to find out if a different dosing schedule of capecitabine combined with neratinib is safer. This different dosing schedule is experimental, meaning the administration schedule of capecitabine and neratinib is not FDA approved for treatment for HER2 positive advanced breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years at signing of informed consent.
* Histologically confirmed MBC, current stage IV.
* Documented HER2 overexpression (immunohistochemistry (IHC) 3+ or gene-amplified tumor with fluorescence in situ hybridization (FISH) ratio of ≥ 2.0.
* For phase Ib, any line of prior treatments is permitted including prior neratinib and capecitabine.
* For phase II, up to 4 prior chemotherapy-based treatments in the metastatic setting are allowed. Patients must have had prior trastuzumab-based therapy. Prior neratinib treatment is not permitted. Prior capecitabine is allowed, if not combined with neratinib.
* Measurable or non-measurable disease is permitted as defined by Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) for phase 1b. For phase 2, patients must have measurable disease as defined in RECIST v1.1.
* Left ventricular ejection fraction (LVEF) ≥50% measured by multiple-gated acquisition scan (MUGA) or echocardiogram (ECHO).
* Eastern Cooperative Oncology Group (ECOG) status of 0 to 1
* Hematologic parameters: white blood cell (WBC) count of > 3000/ul, absolute neutrophil count (ANC) ≥ 1000/ul, platelets ≥ 50,000/ul, hemoglobin ≥ 8.0 g/dl
* Non-hematologic parameters: bilirubin ≤ 1.5 mg/dl, AST/ALT ≤ 3.0 x upper limit of normal (ULN) (≤ 5.0 x ULN if liver metastases are involved)
* Creatinine ≤1.5 mg/dl Patients with "treated and stable" brain lesions of a duration of ≥ 2 months may be enrolled.
* Negative β-human chorionic gonadotropin (hCG) pregnancy test for premenopausal women of reproductive capacity (those who are biologically capable of having children) and for women less than 12 months after menopause.
* Women of childbearing potential must agree and commit to the use of a highly effective method of contraception as determined to be acceptable by the investigator, from the time of informed consent until 28 days after the last dose of the investigational product. Men must agree and commit to use a barrier method of contraception while on treatment and for 3 months after last dose of investigational products.
* Provide written, informed consent to participate in the study and follow the study procedures

Exclusion Criteria:

* Active uncontrolled cardiac disease, including cardiomyopathy, congestive heart failure (New York Heart Association functional classification of ≥2), unstable angina, myocardial infarction within 12 months of enrollment, or ventricular arrhythmia
* Received prior therapy resulting in a cumulative epirubicin dose >900 mg/m2 or cumulative doxorubicin dose >450 mg/m2. If another anthracycline or more than one anthracycline has been used, the cumulative dose must not exceed the equivalent of 450 mg/m^2 doxorubicin.
* Any major surgery ≤28 days prior to the initiation of investigational products, or received anti-cancer therapy (including chemotherapy, biological therapy, hormonal therapy, investigational agents, or other anti-cancer therapy) administered ≤14 days prior to the initiation of investigational products.
* Received radiation therapy ≤14 days prior to initiation of investigational products.
* QTc interval >450 ms for men or 470 ms for women, or known history of QTc prolongation or Torsades de Pointes.
* Active hepatitis B or C
* Active infection or unexplained fever >38.5°C (>101.3°F) within 2 weeks prior to enrollment.
* Significant chronic gastrointestinal disorder with diarrhea as a major symptom (e.g., Crohn's disease, malabsorption, or Grade ≥2 diarrhea of any etiology screening).
* Known dihydropyrimidine dehydrogenase deficiency.
* Known hypersensitivity to 5-fluorouracil or to any component of the investigational products or compounds of similar chemical composition.
* Pregnant patients or currently breast-feeding.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Breast Cancer
Enrollment: 34 (Actual)
Dates: Start 2017-12-13 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 1 year
  If 0 of the 3 patients entered at a dose level experiences a DLT, another 3 patients will be treated at the next higher dose level. If 1 of 3 patients in a cohort experiences a DLT, then up to 3 additional patients will be treated at the same dose level. If none of these 3 additional patients experience a DLT, then the dose will be escalated to the next higher dose level. If > 2 of the initial 3 or 6 patients at a dose level experience a DLT, then the MTD will have been exceeded, and de-escalation is warranted. De-escalation will continue if > 2 of the initial 3 or 6 patients in a dose level cohort experience a DLT. There will be 2 dose de-escalation levels (dose levels -1 and -2) and one dose escalation (dose level +1) as shown in the table below. If < 1 of 6 patients, at that dose level, experience a DLT, then that dose level will be confirmed as the MTD.

CONTACTS AND LOCATIONS:
Overall Officials: Chau Dang, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (10):
- United States (10):
  - Hartford Healthcare Cancer Institute @ Hartford Hospital, Hartford, Connecticut
  - Baptist Alliance - McI, Miami, Florida
  - Memorial Sloan Kettering at Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Lehigh Valley Health Network, Allentown, Pennsylvania

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm